CLINICAL TRIAL: NCT04489290
Title: A Randomised, Double-blind, and Placebo-controlled Post Market Clinical Follow-Up Investigation to Investigate the Clinical Performance of a Medical Device on Clinical Signs and Symptoms, and the Vaginal Environment in Patients With Bacterial Vaginosis
Brief Title: Efficacy and Safety of D005 Vaginal Mousse on Bacterial Vaginosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PepTonic Medical AB (Industry)
Collaborators: Key2Compliance (Industry); CPS Research (Unknown); Scandinavian Development Services AB (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Piva01
Record Dates: First submitted 2020-07-24; First posted 2020-07-28 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Bacterial Vaginosis | Vaginal | Microbiology
Keywords: women's health; bakteriell vaginos
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D005 Vaginal Mousse (Experimental)
  Interventions: Device: D005 Vaginal Mousse
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Device: D005 Vaginal Mousse — D005 Vaginal Mousse is class IIa medical device for treatment of Bacterial Vaginosis.
  Arms: D005 Vaginal Mousse
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomised, double-blind clinical investigation to evaluate the efficacy and safety of D005 vaginal mousse compared to placebo, in women with bacterial vaginosis.

The study will be conducted at one site in Scotland, United Kingdom and at six different sites in Sweden. The study population will consist of approximately 83 female subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability to provide informed consent
2. Female in fertile age
3. Age ≥18 years
4. Bacterial vaginosis, as defined by the following criteria (Amsel criteria):

   1. A fishy odour (i.e., a positive whiff test) of the vaginal discharge with the addition of a drop of potassium hydroxide (KOH)
   2. Presence of clue cells (≥20%)
   3. Off-white (milky or gray), thin, homogeneous discharge
5. Refrain from using any intravaginal products during the investigation period
6. Refrain from sexual intercourse during treatment. Refrain from sexual intercourse or use a condom during rest of the investigation period to Visit 3.

Exclusion Criteria:

1. Hypersensitivity or allergy to the investigational devices or to chemically related products
2. Current use of an intrauterine device.
3. Current pregnancy or intention to become pregnant within 1 month after treatment
4. Antibiotic treatment within 2 weeks before treatment
5. Signs of other infections (such as chlamydia, gonorrhoea, trichomonas, candida, HSV or HPV) requiring specific antibiotic, antifungal or other treatment at screening.
6. Immunosuppression therapy (Allergy medications allowed) at the discretion of the PI
7. Existing or suspected vaginal or cervical cancer or ulcer
8. Unprotected vaginal sex within 24 hours prior to Visit 1
9. Be identified by the Investigator as inappropriate from a medical or compliance perspective to participate in this investigation (e.g. hysterectomised or inability to report daily using smartphone/computer [eDiary]).

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Estimated)
Dates: Start 2021-02-12 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate | 1 to 3 days after last dosing
  Clinical cure at Visit 2, defined as absence of all of the following 3 Amsel criteria:
  1. Off-white (milky or gray), thin, homogeneous discharge.
  2. The presence of clue cells greater than 20% of the total epithelial cells on microscopic examination.
  3. A fishy odour (i.e., a positive whiff test) of the vaginal discharge with the addition of a drop of potassium hydroxide (KOH).

SECONDARY OUTCOMES:
Clinical cure rate | 23 to 28 days after last dosing
  Clinical cure at Visit 3, defined as absence of all of the following 3 Amsel criteria:
  1. Off-white (milky or gray), thin, homogeneous discharge.
  2. The presence of clue cells greater than 20% of the total epithelial cells on microscopic examination.
  3. A fishy odour (i.e., a positive whiff test) of the vaginal discharge with the addition of a drop of KOH.
Modified Hay/Ison <grade III at Visit 2 | 1 to 3 days after last dosing
Modified Hay/Ison <grade III at Visit 3 | 23 to 28 days after last dosing
Clinical cure + Modified Hay/Ison <grade III at Visit 2 | 1 to 3 days after last dosing
Clinical cure + Modified Hay/Ison <grade III at Visit 3 | 23 to 28 days after last dosing
Subject-reported experiences and symptoms of vaginal malodour, discharge or itch during treatment, at Visit 2 | 1 to 3 days after last dosing
  Vaginal malodour, discharge and itch will be graded as the following:
  Vaginal malodour 0 = normal, 1 = mild, 2 = moderate, 3 = severe Discharge 0 = normal, 1 = mild, 2 = moderate Itch 0 = normal, 1 = mild, 2 = moderate, 3 = severe
Subject-reported experiences and symptoms of vaginal malodour, discharge or itch during treatment, at Visit 3 | 23 to 28 days after last dosing
  Vaginal malodour, discharge and itch will be graded as the following:
  Vaginal malodour 0 = normal, 1 = mild, 2 = moderate, 3 = severe Discharge 0 = normal, 1 = mild, 2 = moderate Itch 0 = normal, 1 = mild, 2 = moderate, 3 = severe
pH of the vaginal fluid during treatment | Day 1-7
pH of the vaginal fluid at Visit 2 | 1 to 3 days after last dosing
pH of the vaginal fluid at Visit 3 | 23 to 28 days after last dosing
Absence of clue cells greater than 20 % of the total epithelial cells on microscopic examination at Visit 2 and Visit 3. | 1 to 3 days + 23 to 28 days after last dosing
Total absence of clue cells (0%) of the total epithelial cells on microscopic examination at Visit 2 and Visit 3. | 1 to 3 days + 23 to 28 days after last dosing

CONTACTS AND LOCATIONS:
Locations (9):
- Sweden (8):
  - Ladulaas Kliniska Studier, Borås
  - Hoftekliniken,, Helsingborg
  - Qvinnolivet Praktikertjänst AB, Kungsbacka
  - Hälsomedicinskt Center Barnmorskemottagning, Lomma
  - 2Heal Medical, Stockholm
  - Kvinnokliniken, Danderyds Sjukhus, Stockholm
  - Ondrasek Läkarmottagning, Sundsvall
  - Gynekologisk mottagning Centrum för Obstetrik och gynekologi Norrlands Universitetssjukhus, Umeå
- CPS Research, Glasgow, Scottland, United Kingdom